CLINICAL TRIAL: NCT05786664
Title: A Comprehensive Breast Cancer Survivorship Biorepository
Brief Title: Breast Cancer Survivorship Biorepository
Status: Recruiting | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1B-21-6; NCI-2021-13442 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1B-21-6 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2023-03-15; First posted 2023-03-27 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Invasive Breast Carcinoma
MeSH Terms: interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (survey, biospecimen collection, record review): Patients complete surveys, undergo collection of blood samples, and review of medical records on study.
  Interventions: Procedure: Biospecimen Collection; Other: Electronic Health Record Review; Other: Quality-of-Life Assessment; Other: Survey Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Electronic Health Record Review — Review of records
Other: Quality-of-Life Assessment — Complete quality-of-life questionnaires
  Other Names: Quality of Life Assessment
Other: Survey Administration — Complete surveys

SUMMARY:
This study collects blood samples as well as clinical and self-report data from stage I-III breast cancer survivors to create a biorepository for future use. The creation of this biorepository will allow for future research into links between individual, molecular, and genomic signatures and cancer outcomes.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To create an annotated biorepository with prospectively collected blood samples from breast cancer survivors.

SECONDARY OBJECTIVES:

I. To collect comprehensive data on social determinants of health (e.g., race/ethnicity, acculturation, socioeconomic status, and access to care), environmental exposures (based on zip codes/geocoding), lifestyle (e.g., diet, tobacco use), clinicopathologic characteristics, treatment history, follow-up and current disease status, survivorship-related issues.

II. To establish an efficient process for researchers to utilize the biorepository for breast cancer and survivorship-related studies.

OUTLINE:

Patients complete surveys, undergo collection of blood samples, and review of medical records on study.

ELIGIBILITY:
Inclusion Criteria:

* Women of all racial and ethnic groups 18 years of age or older
* Women with a diagnosis of invasive breast cancer (stages I-III) within the past 7 years
* Women who have completed active treatment for breast cancer (surgery, chemotherapy, HER2-directed therapy and radiation)
* Prior participation on clinical trials is allowed

Exclusion Criteria:

* Current receipt of interventional clinical trial participation
* Stage IV (metastatic) cancer
* Prior history of recurrence (except recurrence following ductal carcinoma in situ)
* Inability to give informed consent
* Unable to speak English, Spanish, Chinese, or Korean

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult women diagnosed with invasive breast cancer (stages I-III) who have completed active treatment.
Sampling Method: Non-Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2022-04-11 (Actual); Primary Completion 2027-04-11 (Estimated); Study Completion 2028-04-11 (Estimated)

PRIMARY OUTCOMES:
Biorepository | 5 years
  Number of biological samples collected and stored (blood)

CONTACTS AND LOCATIONS:
Overall Officials: Bodour Salhia, PhD, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States